CLINICAL TRIAL: NCT06336486
Title: Comparison of the Effectiveness of Pregabalin Therapy on Neuropathic Pain in Patients With Diabetic Polyneuropathy and the Treatments Applied in Patients Receiving Pregabalin and Intermittent Pneumatic Compression Therapy
Brief Title: the Effectiveness of Intermittent Pneumatic Compression on Neuropathic Pain in Patients With Diabetic Polyneuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Busra Gunes (Other)
Responsible Party: Sponsor-Investigator, Busra Gunes, Principal Investigator, Balikesir University
Organization: Balikesir University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BalikesirU-FTR-BG-01
Record Dates: First submitted 2024-03-19; First posted 2024-03-28 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Diabetic Neuropathic Pain
Keywords: Intermittent pneumatic compression; Diabetic Neuropathy; Pain Measurements; Quality of life
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: two groups with a conventional therapy control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intermittent pneumatic compression +pregabalin (Active Comparator): Patients were given an intermittent pneumatic compression program at a pressure of 35 mmhg for 30 min to the lower extremity for 10 days of extreme alternation in our clinic and pregabalin treatment was continued.
  Interventions: Device: intermittent pneumatic compression +pregabalin group
- pregabalin (Other): only pregabalin treatment was continued.
  Interventions: Other: pregabalin group

INTERVENTIONS:
Device: intermittent pneumatic compression +pregabalin group — The investigators divided the patients into two equal groups , some of the patients were given an intermittent pneumatic compression program at a pressure of 35 mmhg for 30 min to the lower extremity for 10 days of extreme alternation in our clinic and pregabalin treatment was continued.
  Arms: intermittent pneumatic compression +pregabalin
Other: pregabalin group — only pregabalin treatment was continued.
  Arms: pregabalin

SUMMARY:
In this study,the effectiveness of intermittent pneumatic compression therapy on neuropathic pain and quality of life in patients with neuropathic pain due to type 2 diabetes was investigated

DETAILED DESCRIPTION:
The investigators conducted our research from 50 patients with type 2 diabetes of 5-20 years, who received pregabalin treatment with diabetic neuropathy with consent form between 40-75 years.The investigators divided the patients into two equal groups , some of the patients were given an intermittent pneumatic compression program at a pressure of 35 mmhg for 30 min to the lower extremity for 10 days of extreme alternation in our clinic and pregabalin treatment was continued,only pregabalin treatment of the other group was continued. VAS, PQAS, LANSS, SF-36 were evaluated.The evaluation was done before the treatment, at the end of the intermittent pneumatic compression treatment(approximately 2 weeks after the start of the treatment) and 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* 5-20 years history of type 2 diabetes
* Between the ages of 40-75
* Body mass 25-40
* Blood pressure 100/60-140/90
* Patient diagnosed with diabetic polyneuropathy
* Use of pregabalin

Exclusion Criteria:

* Connective tissue disease
* Peripheral nerve vasculitis
* Postherpetic neuralgia
* Alcoholic neuropathy
* Autonomic neuropathy
* Chronic renal failure
* Charcot-marie tooth disease

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
The Leeds assessment of neuropathic symptoms and signs(LANSS) | The evaluation was done before the treatment, at the end of the intermittent pneumatic compression treatment(approximately 2 weeks after the start of the treatment) and 3 months later.
  The Leeds Assessment of Neuropathic Symptoms and Signs Pain Scale (LANSS) comprises of a 7-item pain scale, including the sensory descriptors and items for sensory examination.
  Out of the seven items in the Leeds Assessment of Neuropathic Symptoms and Signs Pain Scale (LANSS), five are symptom related and two are examination items. On the LANSS Pain Scale, a score of 12 or more was classified as neuropathic pain, and a score under 12 was classified as nociceptive pain. The intensity of pain at the time of interview was recorded on a 10-cm visual analogue scale (VAS) (0, no pain; 10, unbearable pain).
Pain quality rating scale(PQAS) | The evaluation was done before the treatment, at the end of the intermittent pneumatic compression treatment(approximately 2 weeks after the start of the treatment) and 3 months later.
  The Pain Quality Assessment Scale (PQAS) is an adjusted version of the validated Neuropathic Pain Scale and includes 20 pain qualities and descriptors. PQAS asks respondents to rate the severity of each of 20 pain (quality and spatial) descriptor domains by using 0 to 10 numeric rating scales, in which 0 "no pain" or "not [sensation/item]" and 10 "the most [descriptor] pain sensation imaginable.
Visual Analog Scale(VAS) | The evaluation was done before the treatment, at the end of the intermittent pneumatic compression treatment(approximately 2 weeks after the start of the treatment) and 3 months later.
  . The intensity of pain at the time of interview was recorded on a 10-cm visual analogue scale (VAS) (0, no pain; 10, unbearable pain).

SECONDARY OUTCOMES:
36-Item Short Form Health Survey(SF-36) | The evaluation was done before the treatment, at the end of the intermittent pneumatic compression treatment(approximately 2 weeks after the start of the treatment) and 3 months later.
  The SF-36 measures eight domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health, and has two summary scores (physical and mental).
  For each quality of life domain tested, item scores were coded, summed, and transformed into a scale from 0 (worst) to 100 (best) using the standard SF-36 scoring algorithms. Physical and mental summary component scale scores were also calculated using algorithm described by the developers

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Şahin, Prof., Study Director — Balikesir University
Locations (1):
- Balıkesir University, Balıkesir, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No